CLINICAL TRIAL: NCT04341870
Title: Efficacy of Sarilumab + Azithromycin + Hydroxychloroquine, and Sarilumab Alone, for Adult Patients Hospitalized With Moderate to Severe COVID-19: a Multicenter Open-label 1:1 Randomized Controlled Trial
Brief Title: Study of Immune Modulatory Drugs and Other Treatments in COVID-19 Patients: Sarilumab, Azithromycin, Hydroxychloroquine Trial - CORIMUNO-19 - VIRO
Acronym: CORIMUNO-VIRO
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DSMB recommendation (futility)
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200375-3
Record Dates: First submitted 2020-04-06; First posted 2020-04-10 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: COVID19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — sarilumab; Azithromycin; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Bayesian open labelled randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarilumab + Azithromycin + Hydroxychloroquine (Experimental): Sarilumab combined with Azithromycin and Hydroxychloroquine
  Interventions: Drug: Sarilumab; Drug: Azithromycin; Drug: Hydroxychloroquine
- Sarilumab (Active Comparator): Sarilumab only
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Sarilumab: 400 mg in a 1 hour - I.V. infusion on D1
Drug: Azithromycin — Azithromycin: oral administration, 500mg on D1 then 250mg QD on D2 to D5 (total duration 5 days)
  Arms: Sarilumab + Azithromycin + Hydroxychloroquine
Drug: Hydroxychloroquine — Hydroxychloroquine: oral administration, 600mg QD (200mg TID) from D1 to D10 (total duration 10 days)
  Arms: Sarilumab + Azithromycin + Hydroxychloroquine

SUMMARY:
The overall objective of the study is to determine the therapeutic effect and tolerance of Sarilumab in combination with Azithromycin and Hydroxychloroquine, compared to Sarilumab only, patients with moderate, severe pneumonia associated with Coronavirus disease 2019 (COVID-19). Sarilumab is a human IgG1 monoclonal antibody that binds specifically to both soluble and membrane-bound IL-6Rs (sIL-6Rα and mIL-6Rα) and has been shown to inhibit IL-6-mediated signaling through these receptors. The study has a cohort multiple Randomized Controlled Trials (cmRCT) design. Randomization will occur prior to offering investigational treatments administration to patients enrolled in the CORIMUNO-19 cohort (NCT04324047). Sarilumab+Azithromycin+Hydroxychloroquine, or Sarilumab only will be administered to consenting adult patients hospitalized with COVID-19 either diagnosed with moderate or severe pneumonia requiring no mechanical ventilation. All patients will receive standard of care along with randomized investigational treatments. Outcomes of included patients will be compared between groups as well as with outcomes of patients in the CORIMUNO-19 cohort treated with other immune modulators or standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the CORIMUNO-19 cohort (NCT04324047)
* COVID-19 cases not requiring ICU at admission with moderate or severe pneumopathy according to the WHO Criteria of severity of COVID pneumopathy:

  * Moderate cases: Cases meeting all of the following criteria: [Showing fever and respiratory symptoms with radiological findings of pneumonia] AND [Requiring between 3L/min and 5L/min of oxygen to maintain SpO2>97%] OR
  * Severe cases: Cases meeting any of the following criteria: [Respiratory distress ( ≥ 30 breaths/ min)] OR [Oxygen saturation≤93% at rest in ambient air; or Oxygen saturation ≤97 % with O2 > 5L/min] OR [PaO2/FiO2 ≤ 300mmHg]

Exclusion Criteria:

1. Patients with exclusion criteria to the CORIMUNO-19 cohort.
2. Respiratory failure requiring non invasive or mechanical ventilation
3. Patients requiring intensive care
4. Do-not-resuscitate order (DNR order)
5. Known hypersensitivity to sarilumab or to any of their excipients.
6. Known contra-indication to hydroxychloroquine or chloroquine: including hypersensitivity/allergy, retinopathy, G6PD deficiency and QT prolongation
7. Known contra-indication to azithromycin: including hypersensitivity/allergy and QT prolongation
8. Pregnancy or breastfeeding
9. Current documented bacterial infection.
10. Patient with any of following laboratory results out of the ranges detailed below at screening should be discussed depending of the medication:

    * Absolute neutrophil count (ANC) ≤ 1.0 x 109/L
    * Haemoglobin level: no limitation
    * Platelets (PLT) < 50 G /L
    * SGOT or SGPT > 5N

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-05-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Need for ventilation (including invasive and non invasive ventilation), intensive care or death | 14 days
  Events considered are: need for ventilation (including invasive and non invasive ventilation), transfer to the Intensive Care Unit, death or new do-not-resuscitate (DNR) decision in the absence ventilation and outside ICU.

SECONDARY OUTCOMES:
Early improvement: OMS progression scale <= 5 | 4 days
  WHO progression scale: Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
OMS progression scale | 4, 7 and 14 days
  WHO progression scale: Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Survival | 14, 28 and 90 days
  Overall survival
ICU-free days alive | 14, 28 and 90 days
  Number of ICU-free days alive
Ventilation-free days alive | 14 and 28 days
  Number of ventilation(invasive or non invasive)-free days alive
Hospital-free days alive | 14, 28 and 90 days
  Number of hospital-free days alive
Oxygen therapy-free days alive | 14 and 28 days
  Number of oxygen therapy-free days alive
Time to negative viral excretion | 90 days
  SARS-CoV-2 viral load measurement by rtPCR
Immunophenotyping and multiplex cytokines | 8 days
  Immunophenotyping and multiplex cytokines (blood sample)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - AP-HP Hôpital Avicenne, Bobigny
  - AP-HP Hôpital Ambroise Paré, Boulogne-Billancourt
  - AP-HP Hôpital Beaujon, Clichy
  - AP-HP Hôpital Pitié Salpétrière, Paris
  - AP-HP Hôpital Saint Antoine, Paris

IPD SHARING:
Plan to Share IPD: Undecided